CLINICAL TRIAL: NCT06730880
Title: Detection of Single Nucleotide Polymorphism (SNP) Rs2235371 of IRF6 Gene in Egyptian Patients with Non-Syndromic Cleft Lip and Palate
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Elsharkawy, Dr., Assiut University
Other Study IDs: PCR in Cleft Lip & Palate
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cleft Lip and Cleft Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PCR — Polymerase chain reaction (abbreviated PCR) is a laboratory technique for rapidly producing (amplifying) millions to billions of copies of a specific segment of DNA, which can then be studied in greater detail.

SUMMARY:
The aim of this work is to study the relation between SNP rs2235371 of IRF 6 gene and Non-Syndromic Cleft Lip and Palate in Egyptian Patients in a prospective study

DETAILED DESCRIPTION:
Infants born with facial deformities, such as cleft lip and palate (CL/P), often face lifelong challenges, including communication issues, aesthetic concerns, and difficulty with swallowing, which impact both health and social behavior. Without treatment, these conditions require specialized care and lead to higher rates of morbidity and mortality. Surgeries, including speech and dental interventions, can help manage these conditions from early childhood . CL/P is one of the most common craniofacial birth defects, affecting populations worldwide, with Asian populations experiencing the highest prevalence at 1/500 live births.

Cleft palate (CP) results from incomplete closure of the palate shelves in early prenatal development. Depending on severity, it may range from a minor fissure to a full gap between the mouth and nasal cavity, necessitating surgical repair. CL/P is categorized as syndromic or non-syndromic, with the latter resulting from failure of palatal fusion between 4-12 weeks of embryogenesis, influenced by factors such as single-gene mutations, chromosomal abnormalities, and environmental interactions.

Key genetic mutations linked to CL/P include those in the IRF6, PVRL1, TP63, FGFR1, and TBX22 genes, with IRF6 SNPs being particularly significant . Family history increases risk, while gene-environment interactions, maternal drug use, non-gestational diabetes, and vitamin deficiencies contribute further. A multidisciplinary approach is essential for managing CL/P, supporting children's functional and aesthetic outcomes from birth through adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non-Syndromic Cleft lip or Cleft lip and palate.

Exclusion Criteria:

* Patients with Syndromic CLP.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals diagnosed with cleft lip or cleft lip and palate (CLP). The inclusion criteria are limited to patients with non-syndromic CLP to focus on genetic factors specific to this condition. Patients diagnosed with syndromic CLP, where clefting is associated with other syndromic features or conditions, are excluded to avoid confounding factors and ensure the study's focus remains on non-syndromic cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Study the relation between the presence of SNP rs2235371 and Non-Syndromic CLP | From enrollment to 48 hours after.
  The primary outcome of this study is to investigate the relationship between the presence of the single nucleotide polymorphism (SNP) rs2235371 and the occurrence of non-syndromic cleft lip with or without cleft palate (NSCLP). By analyzing the genetic association between rs2235371 and NSCLP, the research aims to identify potential genetic risk factors contributing to the development of this congenital condition.